CLINICAL TRIAL: NCT05624814
Title: Long-term Psychological Evaluation of Patients With Implanted Spinal Cord Stimulator
Brief Title: Psychological Evaluation After SCS Implantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Other Study IDs: Psico-SCS
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Psychological Disability; Cognitive Impairment; Quality of Life
Keywords: Spinal Cord Stimulation; Psychological Disability; Cognitive Impairment; Quality of Life; Metacognition; Pain and Disability
MeSH Terms: conditions — Cognitive Dysfunction; Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental group: Patients with chronic pain which failed standard therapies and with an implanted Spinal Cord Stimulator
  Interventions: Device: Spinal Cord Stimulation
- Comparison group: Patients with chronic pain following traditional therapies, i.e. pharmacological, psychological, physical and occupational therapies or surgery.
  Interventions: Other: Standard therapies
- Control group: Healthy volunteers matched for age and schooling to those included in the experimental group

INTERVENTIONS:
Device: Spinal Cord Stimulation — Spinal Cord Stimulation consists of the transcutaneous or surgical implantation of different types of electrodes in the epidural space; electrodes are then connected to an Implanted Pulse Generator that generates stimulating currents.
  Groups: Experimental group
Other: Standard therapies — Standard therapies for chronic low back pain are pharmacological, psychological, physical and occupational therapies or surgery.
  Groups: Comparison group

SUMMARY:
Spinal cord stimulation (SCS) is a therapeutic option for patients with chronic low back pain (CLBP) syndrome, when pharmacological, psychological, physical and occupational therapies or surgery fail to reduce symptoms. CLBP is a common disease with several negative consequences on the quality of life, work and activity ability and increased costs to the health-care system. We have therefore designed this observational study to assess global cognitive functioning in three different groups of patients: patients with chronic pain undergoing intervention (experimental group), patients with chronic pain following traditional therapies (comparison group) and healthy participants matched for age and schooling (healthy subjects).

A neuropsychological assessment battery designed to assess global cognitive functioning, behavioral symptomatology, metacognition, quality of life, interoception, pain perception, self-efficacy, and coping styles will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* presence of chronic pain treated with spinal cord stimulation (Experimental Group)
* presence of chronic pain receiving standard therapies (Comparison Group)
* healthy participants matched for age and schooling (Control Group).

Exclusion Criteria:

* consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 consecutive patients (20 per cohort) will be enrolled if they meet the inclusion criteria and no exclusion criteria as per cohort.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Cognitive Functioning - Montreal Cognitive Assessment | At patient's inclusion
  Montreal Cognitive Assessment provides screening of global cognitive functioning; it is composed of 12 subtasks exploring: memory; visuospatial abilities assessed by a clock-drawing task and by copying of a cube; executive functions assessed by means of a brief version of the Trail Making B task, a phonemic fluency task, and a two-item verbal abstraction task; attention, concentration and working memory assessed by means of a sustained attention task (target detection using tapping), a serial subtraction task, and forward and backward span tasks for digits; language assessed by a naming task with low-familiarity animals, repetition of two syntactically complex sentences and the above-mentioned phonemic fluency task; temporal and spatial orientation.
Global Cognitive Functioning - Raven's Colored Progressive Matrices Test | At patient's inclusion
  The Raven's Colored Progressive Matrices Test assesses abstract reasoning abilities with nonverbal material. The test consists of 36 matrices, grouped into 3 sets of increasing difficulty. Each matrix has a missing piece that the subject must choose from six alternatives available. The total score ranges from 0 to 36 and is obtained by summing the number of correct answers.

SECONDARY OUTCOMES:
Metacognition - Memory Assessment Clinics-Questionnaire | At patient's inclusion
  the Memory Assessment Clinics-Questionnaire (MAC-Q) assesses the subjective perception of one's memory performance in daily life compared to the past (for this study, reference will be made before the intervention). It consists of 6 items that assess the subject's ability to remember various information (e.g., phone numbers/postal codes used, location of objects). Each item is measured on a 5-point Likert scale (from ''much better now'' to ''much worse now''). The MAC-Q total score ranges from 7 to 35, with higher scores indicating a greater presence of subjective memory complaints.
Metacognition - Multifactorial Memory Questionnaire | At patient's inclusion
  Multifactorial Memory Questionnaire is a self-administered questionnaire that includes 57 items assessing the three dimensions of metamemory: Satisfaction, Ability, and Strategy.
Metacognition - Adult Executive Functioning Inventory | At patient's inclusion
  The Adult Executive Functioning Inventory (ADEXI; Holst and Thorell, 2018) is a self-administered questionnaire comprising 14 items that assess subjective perceptions of one's inhibition skills and working memory. Each item is measured on a 5-point Likert scale (from ''definitely not true'' to ''definitely true''). The ADEXI total score ranges from 14 to 70, with higher scores indicating greater subjective impairment in the executive domain.
Quality of life | At patient's inclusion
  Quality of Life Assessment Questionnaire (Short Form Health Survey 36, SF-36), which consists of a survey of the patient's health status. It is a 36-item scale, which measures eight domains of health status: physical functioning; physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health. A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. In addition, it is possible to calculate the values of the two synthetic indices, one related to Physical Health (FHH), and the second to Mental Health (MHSI). The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Behavioral Symptomatology - Beck Depression Inventory | At patient's inclusion
  The Beck Depression Inventory (BDI) is a self-report instrument to assess the severity of depression. It consists of 21 items, which assess the presence and intensity of depressive symptoms in the past two weeks, which can be assigned 0 to 3 points. The BDI total score ranges from 0 to 63. The cut-off is equal to 16.
Behavioral Symptomatology - State-Trait Anxiety Inventory | At patient's inclusion
  The State-Trait Anxiety Inventory (Spielberg et al., 1968) is a self-report instrument to assess the severity of anxiety symptoms. It consists of two scales (Y1 and Y2) of 20 items, which assess state anxiety, through questions referring to how the subject feels at the time of questionnaire administration, and trait anxiety, with questions investigating how the subject habitually feels. The scores for the individual scales range from 20 to 80 with a threshold value predictive of anxiety symptomatology placed at 40.
Behavioral Symptomatology - Apathy Evaluation Scale | At patient's inclusion
  The Apathy Evaluation Scale (Marin et al., 1991) is a rating scale to assess apathy consisting of 18 items. The total apathy score ranges from 18 to 72 and is given by the sum of the scores obtained at the items assessing cognitive apathy, behavioral apathy, emotional apathy, and items that are part of the other category. The cut-off is equal to 38.
Pain - Numeric Rating Scale | At patient's inclusion
  The Numeric Rating Scale is an 11-point unidimensional scale that rates pain intensity. The scale consists of a horizontal line, with a range from 0 to 10, corresponding to "no pain" and "worst pain imaginable," respectively. The total score ranges from 0 to 10, with a high score indicating the presence of a greater intensity of pain.
Disability - Roland Morris Disability Questionnaire | At patient's inclusion
  The Roland Morris Disability Questionnaire is a self-administered questionnaire that assesses the patient's disability and limitations in daily life. It consists of 24 items that assess the subject's ability to perform the 24 listed activities. For each item, a score can be given ranging from 0 (that activity is not limited) to 1 (that activity is limited). The total score ranges from 0 to 24, with high scores indicating the presence of a greater disability.
Pain and disability - Pain Catastrophizing Scale | At patient's inclusion
  The Pain Catastrophizing Scale is a scale that assesses catastrophic thinking in relation to pain. It consists of 13 items in which participants are asked to reflect on past painful experiences and to indicate how often certain thoughts and feelings occur when they experience pain. Each item can be given a score ranging from 0 (never) to 4 (always). The total score ranges from 0 to 52, with higher scores indicating a greater presence of catastrophic thoughts.
Resilience, Perceived Self-efficacy, and Coping Styles - Brief Resilience Scale | At patient's inclusion
  The Brief Resilience Scale (BRS) is a self-administered scale that assesses resilience in stressful situations through 6 items on a 5-point Likert scale (1=completely disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=completely agree). The total score ranges from 6 to 30, with higher scores indicating greater resilience in stressful situations.
Resilience, Perceived Self-efficacy, and Coping Styles - Pain Self-Efficacy Questionnaire | At patient's inclusion
  The Pain Self-Efficacy Questionnaire is a questionnaire used to measure perceived self-efficacy with respect to the presence of pain. It consists of 10 items that describe different daily activities (e.g., I can do most housework) or general aspects of life (e.g., I can still accomplish most of my goals). For each item, the subject must indicate how confident he or she feels that can perform these activities despite the presence of pain. The items are measured on a 7-point Likert scale ranging from 0 (not at all confident) to 6 (completely confident). The total score on the questionnaire can range from 0 to 60, with higher scores indicating greater self-efficacy.
Resilience, Perceived Self-efficacy, and Coping Styles - Coping Scale | At patient's inclusion
  The Coping Scale is a self-administered questionnaire that assesses the use of cognitive, emotional, and behavioral strategies in problem situations. The questionnaire consists of 13 items measured on a 4-point Likert scale (1=not at all; 2=little; 3=somewhat; 4=very much). Scores range from 13 to 52, with higher scores indicating greater levels of coping strategies.
Interoception - Heartbeat Detection Task | At patient's inclusion
  Heartbeat Detection Task will be used to investigate interoceptive accuracy. In this task, participants will be asked to count their heartbeats silently only in their minds, without trying to sense their own pulse or heartbeat. They will be asked to wear a wristwatch for objective measurement of heart rate. Three counting phases of 25 sec, 45 sec, and 65 sec durations, interspersed with 30 sec rest, will be carried out and repeated twice. The order of the phases will be randomized. The level of agreement between measured heart rate and reported subjective perception will be considered a relatively reliable characteristic of "interoceptive accuracy."
Interoception - Self Awareness Questionnaire | At patient's inclusion
  The Self Awareness Questionnaire will be used to investigate interoceptive sensitivity. It consists of 35 items measured on a five-point Likert scale (0 = never to 4 = always). The total score is the sum of all items and ranges from 0 to 140. Higher scores indicate higher levels of interoceptive awareness.
Interoceptive awareness | At patient's inclusion
  Interoceptive awareness will be investigated using a self-report measure that assesses the individual perception of the degree of accuracy of perceived interoceptive (cardiac) information. The relationship between objective interoceptive accuracy and subjective assessment of one's interoceptive accuracy is calculated to obtain a metacognitive measure of how the perceived degree of interoceptive accuracy corresponds to objectively measured interoceptive accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared with al researchers after publication, on reasonable scientific request to the Principal Investigator
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study publication
Access Criteria: On reasonable scientific request by email the Principal Investigator